CLINICAL TRIAL: NCT02548585
Title: A Phase 1/2, Randomized, Double-blind, Placebo-controlled, Multiple-ascending-dose Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of MEDI0382 in Overweight and Obese Subjects With a History of Type 2 Diabetes Mellitus
Brief Title: A Multiple-ascending-dose Study to Evaluate the Efficacy, Safety, and Pharmacokinetics (PK) of MEDI0382 in Overweight and Obese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5670C00002
Record Dates: First submitted 2015-09-04; First posted 2015-09-14 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: MEDI0382, diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Placebo (Placebo Comparator): Participants will receive placebo (matched to either 100 micrograms [mcg], or 150 mcg or 200 mcg or 300 mcg of MEDI0382) subcutaneously (SC) once daily from Day 1 to Day 7 (Cohort 1); or Day 1 to Day 11 (Cohort 2); or Day 1 to Day 15 (Cohort 3); or Day 1 to Day 41 (Cohort 4); or Day 1 to Day 22 (Cohort 5); or Day 1 to Day 17 (Cohort 6).
  Interventions: Drug: Placebo
- Cohort 1: MEDI0382 100 mcg (Experimental): Participants will receive MEDI0382 100 mcg SC once daily from Day 1 to Day 7.
  Interventions: Drug: MEDI0382
- Cohort 2: MEDI0382 150 mcg (Experimental): Participants will receive MEDI0382 100 mcg SC once daily for at least 4 days (Day 1 to Day 4) and thereafter, an up titrated dose of MEDI0382 150 mcg SC once daily for 7 days (Day 5 to Day 11).
  Interventions: Drug: MEDI0382
- Cohort 3: MEDI0382 200 mcg (Experimental): Participants will receive MEDI0382 100 mcg SC once daily for at least 4 days (Day 1 to Day 4); thereafter, an up titrated dose of MEDI0382 150 mcg SC once daily for 4 days (Day 5 to Day 8); followed by second up titrated dose of MEDI0382 200 mcg SC once daily for 7 days (Day 9 to Day 15).
  Interventions: Drug: MEDI0382
- Cohort 4: MEDI0382 200 mcg (Experimental): Participants will receive MEDI0382 100 mcg SC once daily for at least 4 days (Day 1 to Day 4); thereafter, an up titrated dose of MEDI0382 150 mcg SC once daily for 4 days (Day 5 to Day 8); followed by second up titrated dose of MEDI0382 200 mcg SC once daily for 4 days (Day 9 to Day 12), then a further MEDI0382 200 mcg SC once daily for 28 days (Day 13 to Day 40) at home-dosing; followed by MEDI0382 200 mcg SC once daily for 1 day in hospital (Day 41).
  Interventions: Drug: MEDI0382
- Cohort 5: MEDI0382 300 mcg (Experimental): Participants will receive MEDI0382 100 mcg SC once daily for at least 5 days (Day 1 to Day 5); thereafter, an up titrated dose of MEDI0382 150 mcg SC once daily for 5 days (Day 6 to Day 10); then a second up titrated dose of MEDI0382 200 mcg SC once daily for 5 days (Day 11 to Day 15); followed by third up titrated dose of MEDI0382 300 mcg SC once daily for 7 days (Day 16 to Day 22).
  Interventions: Drug: MEDI0382
- Cohort 6: MEDI0382 300 mcg (Experimental): Participants will receive MEDI0382 100 mcg SC once daily for at least 5 days (Day 1 to Day 5); thereafter, an up titrated dose of MEDI0382 200 mcg SC once daily for 5 days (Day 6 to Day 10); followed by a second up titrated dose of MEDI0382 300 mcg SC once daily for 7 days (Day 11 to Day 17).
  Interventions: Drug: MEDI0382

INTERVENTIONS:
Drug: MEDI0382 — MEDI0382 administered subcutaneously.
  Arms: Cohort 1: MEDI0382 100 mcg; Cohort 2: MEDI0382 150 mcg; Cohort 3: MEDI0382 200 mcg; Cohort 4: MEDI0382 200 mcg; Cohort 5: MEDI0382 300 mcg; Cohort 6: MEDI0382 300 mcg
Drug: Placebo — Placebo administered subcutaneously.
  Arms: Placebo

SUMMARY:
A Phase 1/2, multiple dose study with 6 cohorts of ascending doses designed to evaluate the efficacy, safety and pharmacokinetics (PK) of MEDI0382 in participants with Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled study designed to evaluate the efficacy, safety, and PK of MEDI0382 administered as multiple daily SC doses to participants with T2DM. Approximately one hundred and seven participants will be enrolled across 6 cohorts. In cohorts 1-3 the participants will be randomized to MEDI0382 or placebo (2:1). In Cohort 4, participants will be randomized to MEDI0382 or placebo (1:1). In cohort 5 and 6 participants will be randomized to MEDI0382 or placebo (3:1).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM
* Must provide written informed consent
* Body mass index greater than (>) 27 and less than (<) 40 kg/m^2, inclusive
* Venous access suitable for multiple cannulations
* Vital signs within normal specified ranges
* Females must be non-lactating and non-childbearing potential
* Males must practice 2 effective contraceptive measures if sexually active

Exclusion Criteria:

* Any concurrent condition that in the opinion of the investigator would interfere with the evaluation of the investigational product
* History or presence of gastrointestinal, renal, or hepatic disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* History of cancer within the last 10 years, with the exception of non-melanoma skin cancer
* Any clinically important illness (except for T2DM), medical/surgical procedure, or trauma within 4 weeks prior to dosing
* Fasting glucose greater than or equal to (>=) 200 mg/dL
* Positive Hepatitis B, Hepatitis C or human immunodeficiency virus test or use of antiretroviral medications at screening.
* Concurrent or previous use of a glucagon-like peptide 1 receptor agonist
* Current or previous use of systemic corticosteroids within the past 28 days prior to screening
* Use of any medicinal products or herbal preparations licensed for control of body weight or appetite is prohibited.
* Known or suspected history of alcohol or drug abuse within the past 3 years.
* Positive drug screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stumvoll, Principal Investigator — Universitätsklinikum Leipzig
Locations (11):
- Germany (11):
  - Research Site, Berlin
  - Research Site, Erfurt
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Neu-Ulm
  - Research Site, Neuss

REFERENCES:
- [Derived] Bosch R, Petrone M, Arends R, Vicini P, Sijbrands EJG, Hoefman S, Snelder N. Characterisation of cotadutide's dual GLP-1/glucagon receptor agonistic effects on glycaemic control using an in vivo human glucose regulation quantitative systems pharmacology model. Br J Pharmacol. 2024 Jun;181(12):1874-1885. doi: 10.1111/bph.16336. Epub 2024 Feb 25. PMID 38403793
- [Derived] Ambery P, Parker VE, Stumvoll M, Posch MG, Heise T, Plum-Moerschel L, Tsai LF, Robertson D, Jain M, Petrone M, Rondinone C, Hirshberg B, Jermutus L. MEDI0382, a GLP-1 and glucagon receptor dual agonist, in obese or overweight patients with type 2 diabetes: a randomised, controlled, double-blind, ascending dose and phase 2a study. Lancet. 2018 Jun 30;391(10140):2607-2618. doi: 10.1016/S0140-6736(18)30726-8. Epub 2018 Jun 23. PMID 29945727
- See also: D5670C00002 Protocol_Amendment_8-redacted_correct_PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3139&filename=D5670C00002-Protocol_Amendment_8-redacted_correct_PDF-A.pdf
- See also: Statistical_Analysis_Plan_MEDI0382_D5670C00002_Redacted_PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3139&filename=Statistical_Analysis_Plan_MEDI0382_D5670C00002_Redacted_PDF-A.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 09 Dec 2015 to 24 Feb 2017 in Germany.
Pre-assignment Details: A total of 422 participants were screened, of which 113 participants were randomized in the study.
Groups:
- Placebo: Participants received placebo (matched to either 100 micrograms [mcg], or 150 mcg or 200 mcg or 300 mcg of MEDI0382) subcutaneously (SC) once daily from Day 1 to Day 7 (Cohort 1); or Day 1 to Day 11 (Cohort 2); or Day 1 to Day 15 (Cohort 3); or Day 1 to Day 41 (Cohort 4); or Day 1 to Day 22 (Cohort 5); or Day 1 to Day 17 (Cohort 6).
- Cohort 1: MEDI0382 100 mcg: Participants received MEDI0382 100 mcg SC once daily from Day 1 to Day 7.
- Cohort 2: MEDI0382 150 mcg: Participants received MEDI0382 100 mcg SC once daily for at least 4 days (Day 1 to Day 4) and thereafter, an up titrated dose of MEDI0382 150 mcg SC once daily for 7 days (Day 5 to Day 11).
- Cohort 3: MEDI0382 200 mcg: Participants received MEDI0382 100 mcg SC once daily for at least 4 days (Day 1 to Day 4); thereafter, an up titrated dose of MEDI0382 150 mcg SC once daily for 4 days (Day 5 to Day 8); followed by second up titrated dose of MEDI0382 200 mcg SC once daily for 7 days (Day 9 to Day 15).
- Cohort 4: MEDI0382 200 mcg: Participants received MEDI0382 100 mcg SC once daily for at least 4 days (Day 1 to Day 4); thereafter, an up titrated dose of MEDI0382 150 mcg SC once daily for 4 days (Day 5 to Day 8); followed by second up titrated dose of MEDI0382 200 mcg SC once daily for 4 days (Day 9 to Day 12), then a further MEDI0382 200 mcg SC once daily for 28 days (Day 13 to Day 40) at home-dosing; followed by MEDI0382 200 mcg SC once daily for 1 day in hospital (Day 41).
- Cohort 5: MEDI0382 300 mcg: Participants received MEDI0382 100 mcg SC once daily for at least 5 days (Day 1 to Day 5); thereafter, an up titrated dose of MEDI0382 150 mcg SC once daily for 5 days (Day 6 to Day 10); then a second up titrated dose of MEDI0382 200 mcg SC once daily for 5 days (Day 11 to Day 15); followed by third up titrated dose of MEDI0382 300 mcg SC once daily for 7 days (Day 16 to Day 22).
- Cohort 6: MEDI0382 300 mcg: Participants received MEDI0382 100 mcg SC once daily for at least 5 days (Day 1 to Day 5); thereafter, an up titrated dose of MEDI0382 200 mcg SC once daily for 5 days (Day 6 to Day 10); followed by a second up titrated dose of MEDI0382 300 mcg SC once daily for 7 days (Day 11 to Day 17).
Period: Overall Study
Arm/Group | Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: MEDI0382 150 mcg | Cohort 3: MEDI0382 200 mcg | Cohort 4: MEDI0382 200 mcg | Cohort 5: MEDI0382 300 mcg | Cohort 6: MEDI0382 300 mcg
Started | 45 | 6 | 6 | 7 | 25 | 12 | 12
Treated | 45 | 6 | 6 | 7 | 25 | 11 | 12
Completed | 43 | 6 | 6 | 5 | 22 | 10 | 11
Not Completed | 2 | 0 | 0 | 2 | 3 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 2 | 3 | 0 | 1
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: As-treated Population (ATP) included all participants who received any study drug and analyzed according to the treatment they actually received.
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: MEDI0382 150 mcg | Cohort 3: MEDI0382 200 mcg | Cohort 4: MEDI0382 200 mcg | Cohort 5: MEDI0382 300 mcg | Cohort 6: MEDI0382 300 mcg | TOTAL
Number analyzed (Participants) | 45 | 6 | 6 | 7 | 25 | 11 | 12 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (6.0) | 62.5 (2.9) | 60.2 (4.2) | 57.0 (4.9) | 56.0 (7.2) | 54.8 (6.8) | 54.6 (6.5) | 56.9 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 1 | 4 | 2 | 12 | 4 | 3 | 44
  Male | 27 | 5 | 2 | 5 | 13 | 7 | 9 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 45 | 6 | 6 | 7 | 25 | 11 | 12 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 44 | 6 | 6 | 7 | 25 | 11 | 12 | 111
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Mixed-meal Test (MMT) Glucose Area Under the Concentration-time Curve From Time 0 to 4 Hours to the End of Treatment (EOT) (Cohort 4)
Description: Mixed-meal test involved consumption of a standardized meal (nutritional supplement containing the components of fat, carbohydrate and protein, which make up a standard MMT) within 5 minutes, and timed serial blood samples were obtained for measurement of glucose and parameters related to glucose metabolism just before and 4 hours (hrs) after consumption of the standardized meal (with no additional food intake during this time).
Time Frame: 0 minutes before; and 15, 30, 45, 60, 90, 120, 180, and 240 minutes post standardized meal intake (SMI) on Baseline (Day -1) and EOT (Day 41)
Population: Pharmacodynamic (PD) population included all participants who received at least 1 dose of study drug and had at least 1 post-MMT PD blood sample.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Cohort 4: Placebo: Participants received placebo (matched to MEDI0382 100 mcg) SC once daily for at least 4 days (Day 1 to Day 4); thereafter, an up titrated dose of placebo (matched to MEDI0382 150 mcg) SC once daily for 4 days (Day 5 to Day 8); followed by second up titrated dose of placebo (matched to MEDI0382 200 mcg) SC once daily for 4 days (Day 9 to Day 12), then a further placebo (matched to MEDI0382 200 mcg) SC once daily for 28 days (Day 13 to Day 40) at home-dosing; followed by placebo (matched to MEDI0382 200 mcg) SC once daily for 1 day in hospital (Day 41).
Arm/Group | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg
Number analyzed (Participants) | 26 | 25
Percent change | -9.24 (12.30) | -33.81 (18.62)
Statistical Analysis 1: Comparison: Cohort 4: Placebo vs Cohort 4: MEDI0382 200 mcg; Test type: Superiority; p < 0.0001, ANCOVA; p-value was based on pairwise comparison using analysis of covariance (ANCOVA) adjusted by baseline value

2. Primary Outcome: Change From Baseline in Body Weight to the EOT (Cohort 4)
Time Frame: Baseline (Day 1) and EOT (Day 42)
Population: Intent-to-treat (ITT) population included all participants who were randomized and received any study drug and analyzed according to the initial randomization.
Measure: Mean (Standard Deviation); unit: Kilograms (Kg)
Arm/Group | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg
Number analyzed (Participants) | 26 | 25
Kilograms (Kg) | -1.71 (2.10) | -3.83 (2.09)
Statistical Analysis 1: Comparison: Cohort 4: Placebo vs Cohort 4: MEDI0382 200 mcg; Test type: Superiority; p = 0.0008, ANCOVA; p-value was based on pairwise comparison using ANCOVA adjusted by baseline value

3. Secondary Outcome: Percent Change From Baseline in MMT Glucose AUC0-4h to the EOT (Cohorts 1, 2, 3, 5, and 6)
Description: Mixed-meal test involved consumption of a standardized meal (nutritional supplement containing the components of fat, carbohydrate and protein, which make up a standard MMT) within 5 minutes, and timed serial blood samples were obtained for measurement of glucose and parameters related to glucose metabolism just before and 4 hrs after consumption of the standardized meal (with no additional food intake during this time).
Time Frame: 0 minutes before; and 15, 30, 45, 60, 90, 120, 180, and 240 minutes post SMI on Baseline (Day -1) and EOT (Day 7 for Cohort 1; Day 11 for Cohort 2; Day 15 for Cohort 3; Day 22 for Cohort 5; and Day 17 for Cohort 6)
Population: PD population included all participants who received at least 1 dose of study drug and had at least 1 post-MMT PD blood sample.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Cohort 1: Placebo: Participants received placebo matched to (MEDI0382 100 mcg) SC once daily from Day 1 to Day 7.
- Cohort 2: Placebo: Participants received placebo (matched to MEDI0382 100 mcg) SC once daily for at least 4 days (Day 1 to Day 4) and thereafter, an up titrated dose of placebo (matched to MEDI0382 150 mcg) SC once daily for 7 days (Day 5 to Day 11).
- Cohort 3: Placebo: Participants received placebo (matched to MEDI0382 100 mcg) SC once daily for at least 4 days (Day 1 to Day 4); thereafter, an up titrated dose of placebo (matched to MEDI0382 150 mcg) SC once daily for 4 days (Day 5 to Day 8); followed by second up titrated dose of placebo (matched to MEDI0382 200 mcg) SC once daily for 7 days (Day 9 to Day 15).
- Cohort 5: Placebo: Participants received placebo (matched to MEDI0382 100 mcg ) SC once daily for at least 5 days (Day 1 to Day 5); thereafter, an up titrated dose of placebo (matched to MEDI0382 150 mcg) SC once daily for 5 days (Day 6 to Day 10); then a second up titrated dose of placebo (matched to MEDI0382 200 mcg) SC once daily for 5 days (Day 11 to Day 15); followed by third up titrated dose of placebo (matched to MEDI0382 300 mcg) SC once daily for 7 days (Day 16 to Day 22).
- Cohort 6: Placebo: Participants received placebo (matched to MEDI0382 100 mcg) SC once daily for at least 5 days (Day 1 to Day 5); thereafter, an up titrated dose of placebo (matched to MEDI0382 200 mcg) SC once daily for 5 days (Day 6 to Day 10); followed by a second up titrated dose of placebo (matched to MEDI0382 300 mcg) SC once daily for 7 days (Day 11 to Day 17).
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 5 | 11 | 5 | 12
Percent change | -14.60 (5.56) | -41.80 (11.07) | -15.07 (13.46) | -36.73 (10.09) | -0.47 (15.16) | -39.58 (5.27) | -14.52 (8.12) | -41.66 (9.97) | -4.80 (3.45) | -38.19 (12.51)

4. Secondary Outcome: Change From Baseline in Body Weight to the EOT (Cohorts 1, 2, 3, 5, and 6)
Time Frame: Cohort 1: Baseline (Day 1) to EOT (Day 8); Cohort 2: Baseline (Day 1) to EOT (Day 12); Cohort 3: Baseline (Day 1) to EOT (Day 16); Cohort 5: Baseline (Day 1) to EOT (Day 22); Cohort 6: Baseline (Day 1) to EOT (Day 17)
Population: ITT population included all participants who were randomized and received any study drug and analyzed according to the initial randomization. Participants who did not complete the treatment were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 5 | 11 | 5 | 12
Kg | -1.20 (0.44) | -2.32 (1.29) | -1.00 (1.13) | -1.52 (0.57) | -2.90 (1.05) | -4.63 (1.98) | -0.98 (2.12) | -3.26 (1.99) | -0.94 (3.09) | -2.04 (1.52)

5. Secondary Outcome: Percent Change From Baseline in Hemoglobin A1c (HbA1c) to the EOT (Cohorts 4, 5, and 6)
Time Frame: Cohort 4: Baseline (Day -2) to EOT (Day 42); Cohort 5: Baseline (Day -2) to EOT (Day 22); Cohort 6: Baseline (Day -2) to EOT (Day 17)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 26 | 25 | 5 | 11 | 5 | 12
Percent change | -0.58 (0.30) | -0.92 (0.41) | -0.10 (0.29) | -0.55 (0.35) | -0.18 (0.19) | -0.42 (0.27)

6. Secondary Outcome: Change From Baseline in Fructosamine to the EOT (Cohorts 4, 5, and 6)
Time Frame: Cohort 4: Baseline (Day -2) to EOT (Day 41); Cohort 5: Baseline (Day -2) to EOT (Day 22); Cohort 6: Baseline (Day -2) to EOT (Day 17)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 26 | 25 | 5 | 11 | 5 | 12
micromol/L | -33.7 (44.6) | -67.9 (44.4) | -27.8 (25.8) | -47.4 (15.7) | -48.8 (43.7) | -47.5 (55.3)

7. Secondary Outcome: Change From Baseline in Fasting Glucose Prior to MMT to the EOT (Cohorts 1, 2, 3, 4, 5, and 6)
Description: as for outcome 3
Time Frame: Cohort 1: Baseline (Day-1) to EOT (Day7); Cohort 2: Baseline (Day-1) to EOT (Day11); Cohort 3: Baseline (Day-1) to EOT (Day15); Cohort 4: Baseline (Day-1) to EOT (Day41); Cohort 5: Baseline (Day-1) to EOT (Day22); Cohort 6: Baseline (Day-1) to EOT (Day17)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25 | 5 | 11 | 5 | 12
mg/dL | -32.44 (17.19) | -74.48 (24.59) | -49.86 (23.24) | -54.06 (19.51) | -4.20 (33.73) | -63.67 (11.93) | -18.52 (18.88) | -50.62 (33.61) | -32.08 (17.49) | -54.42 (19.75) | -16.58 (12.45) | -55.21 (31.13)

8. Secondary Outcome: Percent Change From Baseline in Glucose Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC0-24h) After MMT to the EOT (Cohorts 1, 2, 3, 4, 5, and 6)
Description: as for outcome 3
Time Frame: 0 minutes before; and 15, 30, 45, 60, 90, 120, 180, 240 minutes, and 24 hrs post SMI on Baseline (Day -1) and EOT (Day 7 for Cohort 1; Day 11 for Cohort 2; Day 15 for Cohort 3; Day 41 for Cohort 4; Day 22 for Cohort 5; and Day 17 for Cohort 6)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25 | 5 | 11 | 5 | 12
Percent change | -21.80 (1.41) | -28.34 (13.52) | 0.80 (39.55) | -29.32 (17.24) | -13.80 (15.95) | -27.07 (10.82) | -1.06 (11.47) | -13.50 (18.19) | -4.20 (28.58) | -34.51 (11.25) | -10.10 (14.69) | -26.95 (9.45)

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) is any unfavourable and unintended sign, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. Serious adverse events (SAE) is any AE that resulted in death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, life-threatening, a congenital anomaly/birth defect, or an important medical event. TEAEs and TESAEs are defined as AEs and SAEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 28 days after the last study dose of each cohort (approximately 60 days).
Time Frame: From Day 1 to follow-up period (28 days after the last study dose for each cohort [approximately 60 days])
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25 | 5 | 11 | 5 | 12
Participants
  TEAEs | 2 | 6 | 3 | 5 | 3 | 7 | 23 | 22 | 4 | 10 | 2 | 10
  TESAEs | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Abnormal Vital Signs and Physical Examination Reported as TEAEs
Description: TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 28 days after the last study dose of each cohort (approximately 60 days). Number of participants with TEAEs related to vital signs and physical examination abnormalities were reported.
Time Frame: From Day 1 to follow-up period (28 days after the last study dose for each cohort [approximately 60 days])
Population: ATP included all participants who received any study drug and analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25 | 5 | 11 | 5 | 12
Participants
  Blood Pressure increased | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Blood pressure systolic increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Blood pressure diastolic increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Physical Examinations | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Abnormal 12 Lead Electrocardiogram (ECG) Reported as TEAEs
Description: TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 28 days after the last study dose of each cohort (approximately 60 days). Number of participants with TEAEs related to ECG abnormalities were reported.
Time Frame: From Day 1 to follow-up period (28 days after the last study dose for each cohort [approximately 60 days])
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25 | 5 | 11 | 5 | 12
Participants
  Arrhythmia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Atrial fibrillation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Atrioventricular block first degree | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Atrioventricular block second degree | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Electrocardiogram ST segment depression | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Extrasystoles | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sinus tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Supraventricular extrasystoles | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Supraventricular tachycardia | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Tachycardia | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Ventricular extrasystoles | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Ventricular tachycardia | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Reported as TEAEs
Description: TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 28 days after the last study dose of each cohort (approximately 60 days). Number of participants with TEAEs related to laboratory abnormalities were reported.
Time Frame: From Day 1 to follow-up period (28 days after the last study dose for each cohort [approximately 60 days])
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25 | 5 | 11 | 5 | 12
Participants
  Lipase increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
  Hypokalemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  C-reactive protein increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Chromaturia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

13. Secondary Outcome: Number of Participants With Any Suicidal Ideation as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Score (Cohorts 4, 5, and 6)
Description: The C-SSRS is an interview-based rating scale to systematically assess suicidal ideation and suicidal behaviour of participants. Yes/No responses are mapped to C-SSRS to assess whether participant experienced suicidal behaviour and suicidal ideation. Suicidal behaviour questions includes preparatory acts or behaviour, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation questions includes wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intent to act, active suicidal ideation with some intent to act (without specific plan), and active suicidal ideation with specific plan and intent. Participants with yes response to any category for suicidal ideation were reported below.
Time Frame: Cohort 4: Day -1, and Days 13, 20, 27, 34, and 40; Cohort 5: Day -1 and Day 7-14 post last dose of MEDI0382 (approximately 36 days); Cohort 6: Day -1 and Day 7-14 post last dose of MEDI0382 (approximately 31 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 26 | 25 | 5 | 11 | 5 | 12
Participants
  Day -1 | 1 | 4 | 0 | 2 | 0 | 2
  Day 13: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 13 | 1 | 0 |  |  |  |
  Day 20: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 20 | 0 | 0 |  |  |  |
  Day 27: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 27 | 0 | 0 |  |  |  |
  Day 34: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 34 | 0 | 0 |  |  |  |
  Day 40: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 40 | 0 | 0 |  |  |  |
  Days 7-14 post last dose of MEDI0382: number analyzed (Participants) | 0 | 0 | 5 | 11 | 5 | 12
  Days 7-14 post last dose of MEDI0382 |  |  | 0 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Any Suicidal Behaviour as Assessed by C-SSRS Score (Cohorts 4, 5, and 6)
Description: The C-SSRS is an interview-based rating scale to systematically assess suicidal ideation and suicidal behaviour of participants. Yes/No responses are mapped to C-SSRS to assess whether participant experienced suicidal behaviour and suicidal ideation. Suicidal behaviour questions includes preparatory acts or behaviour, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation questions includes wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intent to act, active suicidal ideation with some intent to act (without specific plan), and active suicidal ideation with specific plan and intent. Participants with yes response to any category for suicidal behaviour were reported below.
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 26 | 25 | 5 | 11 | 5 | 12
Participants
  Day -1 | 2 | 2 | 0 | 1 | 0 | 1
  Day 13: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 13 | 1 | 0 |  |  |  |
  Day 20: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 20 | 0 | 0 |  |  |  |
  Day 27: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 27 | 0 | 0 |  |  |  |
  Day 34: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 34 | 0 | 0 |  |  |  |
  Day 40: number analyzed (Participants) | 26 | 25 | 0 | 0 | 0 | 0
  Day 40 | 0 | 0 |  |  |  |
  Days 7-14 post last dose of MEDI0382: number analyzed (Participants) | 0 | 0 | 5 | 11 | 5 | 12
  Days 7-14 post last dose of MEDI0382 |  |  | 0 | 0 | 0 | 0

15. Secondary Outcome: Terminal Elimination Half Life (t1/2) of MEDI0382 (Cohorts 1, 2, and 3)
Description: Terminal elimination half Life is the time measured for the plasma concentration of MEDI0382 to decrease by one half.
Time Frame: Cohort (C) 1 (Day [D] 1 and [&] D7), C2 (D5 & D11), and C3 (D9 & D15): pre-dose & 0.5, 1, 2, 4, 6, 8, 12, 24 hr post dose; and additional 48 hr post C1D7, C2D11, C3D15 dose
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of study drug and had at least one PK sample taken that was above the lower limit of quantitation.
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Cohort 1: MEDI0382 100 mcg | Cohort 2: MEDI0382 150 mcg | Cohort 3: MEDI0382 200 mcg
Number analyzed (Participants) | 6 | 6 | 7
hr
  Day 1: number analyzed (Participants) | 1 | 0 | 0
  Day 1 | 8.5 [NA to NA] — 95% confidence interval (CI) was not reported as only one participant was evaluable for the specified time point. |  |
  Day 5: number analyzed (Participants) | 0 | 2 | 0
  Day 5 |  | 10.3 [7.8 to 13.5] |
  Day 7: number analyzed (Participants) | 3 | 0 | 0
  Day 7 | 11.7 [5.5 to 25.1] |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 1
  Day 9 |  |  | 8.3 [NA to NA] — 95% CI was not reported as only one participant was evaluable for the specified time point.
  Day 11: number analyzed (Participants) | 0 | 6 | 0
  Day 11 |  | 11.3 [5.9 to 21.7] |
  Day 15: number analyzed (Participants) | 0 | 0 | 5
  Day 15 |  |  | 11.3 [8.2 to 15.5]

16. Secondary Outcome: Accumulation Ratio (Rac) of MEDI0382 (Cohorts 1, 2, and 3)
Description: Accumulation ratio was calculated as, Rac obtained from area under the curve from time zero to end of dosing interval (AUC[0-tau]) of Nth day divided by AUC(0-tau) of Day 1.
Time Frame: C1 (D1 & D7), C2 (D5 & D11), and C3 (D9 & D15): pre-dose & 0.5, 1, 2, 4, 6, 8, 12, 24 hr post dose; and additional 48 hr post C1D7, C2D11, C3D15 dose
Population: PK population included all participants who received at least 1 dose of study drug and had at least one PK sample taken that was above the lower limit of quantitation.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1: MEDI0382 100 mcg | Cohort 2: MEDI0382 150 mcg | Cohort 3: MEDI0382 200 mcg
Number analyzed (Participants) | 6 | 6 | 7
Ratio
  Day 1: number analyzed (Participants) | 6 | 0 | 0
  Day 1 | NA [NA to NA] — Data is not applicable since accumulation ratio, as described by the formula could not be derived for Cohort 1 Day 1. |  |
  Day 5: number analyzed (Participants) | 0 | 6 | 0
  Day 5 |  | NA [NA to NA] — Data is not applicable since accumulation ratio, as described by the formula could not be derived for Cohort 2 Day 5. |
  Day 7: number analyzed (Participants) | 6 | 0 | 0
  Day 7 | 1.3 [1.1 to 1.5] |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 6
  Day 9 |  |  | NA [NA to NA] — Data is not applicable since accumulation ratio, as described by the formula could not be derived for Cohort 3 Day 9.
  Day 11: number analyzed (Participants) | 0 | 6 | 0
  Day 11 |  | 1.1 [0.9 to 1.8] |
  Day 15: number analyzed (Participants) | 0 | 0 | 5
  Day 15 |  |  | 1.3 [1.1 to 1.5]

17. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to End of Dosing Interval (AUC[0-tau]) of MEDI0382 (Cohorts 1, 2, 3, 4, 5, and 6)
Time Frame: C1 (D1 & D7), C2 (D5 & D11), and C3 (D9 & D15): pre-dose & 0.5, 1, 2, 4, 6, 8, 12, 24 hr post dose and 48 hr post dose for C1D7, C2D11, C3D15; C4 (D9 & D41), C5 (D16 & D22), and C6 (D11 & D17): pre-dose & 0.5, 1, 2, 4, 6, 8, 12, 24 hr post dose
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Cohort 1: MEDI0382 100 mcg | Cohort 2: MEDI0382 150 mcg | Cohort 3: MEDI0382 200 mcg | Cohort 4: MEDI0382 200 mcg | Cohort 5: MEDI0382 300 mcg | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 6 | 6 | 7 | 25 | 11 | 12
ng*hr/mL
  Day 1: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
  Day 1 | 82.21 [44.56 to 151.69] |  |  |  |  |
  Day 5: number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 0
  Day 5 |  | 174.58 [87.41 to 348.67] |  |  |  |
  Day 7: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
  Day 7 | 107.01 [54.10 to 211.64] |  |  |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 4 | 23 | 0 | 0
  Day 9 |  |  | 194.78 [146.17 to 259.56] | 164.05 [42.67 to 630.76] |  |
  Day 11: number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 11
  Day 11 |  | 157.31 [82.45 to 421.12] |  |  |  | 275.29 [169.33 to 447.48]
  Day 15: number analyzed (Participants) | 0 | 0 | 5 | 0 | 0 | 0
  Day 15 |  |  | 195.40 [89.8 to 425.17] |  |  |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 0
  Day 16 |  |  |  |  | 261.90 [166.58 to 411.74] |
  Day 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  Day 17 |  |  |  |  |  | 246.06 [130.34 to 464.51]
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0
  Day 22 |  |  |  |  | 254.35 [196.10 to 329.9] |
  Day 41: number analyzed (Participants) | 0 | 0 | 0 | 22 | 0 | 0
  Day 41 |  |  |  | 199.10 [84.57 to 468.75] |  |

18. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - Inf)] of MEDI0382 (Cohorts 1, 2, 3, 4, 5, and 6)
Time Frame: C1 (D1 & D7), C2 (D5 & D11), and C3 (D9 & D15): pre-dose & 0.5, 1, 2, 4, 6, 8, 12, 24 hr post dose and additional 48 hr post dose for C1D7, C2D11, C3D15; C4 (D9 & D41), C5 (D16 & D22), and C6 (D11 & D17): pre-dose & 0.5, 1, 2, 4, 6, 8, 12, 24 hr post dose
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Cohort 1: MEDI0382 100 mcg | Cohort 2: MEDI0382 150 mcg | Cohort 3: MEDI0382 200 mcg | Cohort 4: MEDI0382 200 mcg | Cohort 5: MEDI0382 300 mcg | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 6 | 6 | 7 | 25 | 11 | 12
ng*hr/mL
  Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Day 1 | 103.46 [NA to NA] — 95% CI data not applicable as only one participant was evaluable for this time point. |  |  |  |  |
  Day 5: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0
  Day 5 |  | 207.15 [11.98 to 3580.41] |  |  |  |
  Day 7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0
  Day 7 | 184.68 [107.76 to 316.51] |  |  |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 1 | 13 | 0 | 0
  Day 9 |  |  | 242.60 [NA to NA] — 95% CI data not applicable as only one participant was evaluable for this time point. | 238.22 [80.99 to 700.67] |  |
  Day 11: number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 0
  Day 11 |  | 215.80 [112.90 to 412.47] |  |  |  |
  Day 15: number analyzed (Participants) | 0 | 0 | 5 | 0 | 0 | 0
  Day 15 |  |  | 271.84 [119.33 to 619.24] |  |  |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0
  Day 16 |  |  |  |  | 317.93 [182.24 to 554.64] |
  Day 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4
  Day 17 |  |  |  |  |  | 327.28 [249.98 to 428.49]
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0
  Day 22 |  |  |  |  | 294.60 [172.52 to 503.05] |
  Day 41: number analyzed (Participants) | 0 | 0 | 0 | 11 | 0 | 0
  Day 41 |  |  |  | 262.17 [99.79 to 688.77] |  |

19. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MEDI0382 (Cohorts 1, 2, 3, 4, 5, and 6)
Time Frame: as for outcome 18
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1: MEDI0382 100 mcg | Cohort 2: MEDI0382 150 mcg | Cohort 3: MEDI0382 200 mcg | Cohort 4: MEDI0382 200 mcg | Cohort 5: MEDI0382 300 mcg | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 6 | 6 | 7 | 25 | 11 | 12
ng/mL
  Day 1: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
  Day 1 | 4.97 [0.33 to 7.41] |  |  |  |  |
  Day 5: number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 0
  Day 5 |  | 9.66 [4.68 to 19.95] |  |  |  |
  Day 7: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
  Day 7 | 6.26 [3.36 to 11.67] |  |  |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 6 | 23 | 0 | 0
  Day 9 |  |  | 10.57 [6.33 to 17.66] | 11.64 [3.16 to 42.94] |  |
  Day 11: number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 11
  Day 11 |  | 9.57 [4.63 to 19.79] |  |  |  | 13.69 [5.73 to 32.71]
  Day 15: number analyzed (Participants) | 0 | 0 | 5 | 0 | 0 | 0
  Day 15 |  |  | 10.97 [4.62 to 26.06] |  |  |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 0
  Day 16 |  |  |  |  | 17.65 [8.82 to 35.29] |
  Day 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  Day 17 |  |  |  |  |  | 15.55 [7.55 to 32.01]
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0
  Day 22 |  |  |  |  | 15.77 [10.02 to 24.8] |
  Day 41: number analyzed (Participants) | 0 | 0 | 0 | 22 | 0 | 0
  Day 41 |  |  |  | 13.42 [4.77 to 37.75] |  |

20. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of MEDI0382 (Cohorts 1, 2, 3, 4, 5, and 6)
Time Frame: as for outcome 18
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1: MEDI0382 100 mcg | Cohort 2: MEDI0382 150 mcg | Cohort 3: MEDI0382 200 mcg | Cohort 4: MEDI0382 200 mcg | Cohort 5: MEDI0382 300 mcg | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 6 | 6 | 7 | 25 | 11 | 12
ng/mL
  Day 1: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
  Day 1 | 0.705 [0.33 to 1.49] |  |  |  |  |
  Day 5: number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 0
  Day 5 |  | 2.685 [1.06 to 6.79] |  |  |  |
  Day 7: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
  Day 7 | 2.372 [1.18 to 4.78] |  |  |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 6 | 23 | 0 | 0
  Day 9 |  |  | 3.521 [2.16 to 5.75] | 2.635 [0.79 to 8.83] |  |
  Day 11: number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 11
  Day 11 |  | 3.59 [1.62 to 7.94] |  |  |  | 3.586 [1.45 to 8.88]
  Day 15: number analyzed (Participants) | 0 | 0 | 5 | 0 | 0 | 0
  Day 15 |  |  | 4.973 [2.24 to 11.05] |  |  |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 0
  Day 16 |  |  |  |  | 4.062 [1.68 to 9.84] |
  Day 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  Day 17 |  |  |  |  |  | 4.766 [2.74 to 8.3]
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0
  Day 22 |  |  |  |  | 5.21 [1.97 to 13.81] |
  Day 41: number analyzed (Participants) | 0 | 0 | 0 | 22 | 0 | 0
  Day 41 |  |  |  | 3.38 [1.03 to 11.04] |  |

21. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of MEDI0382 (Cohorts 1, 2, 3, 4, 5, and 6)
Time Frame: as for outcome 18
Population: as for outcome 16
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 1: MEDI0382 100 mcg | Cohort 2: MEDI0382 150 mcg | Cohort 3: MEDI0382 200 mcg | Cohort 4: MEDI0382 200 mcg | Cohort 5: MEDI0382 300 mcg | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 6 | 6 | 7 | 25 | 11 | 12
hr
  Day 1: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
  Day 1 | 8 [6 to 8] |  |  |  |  |
  Day 5: number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 0
  Day 5 |  | 6 [4 to 8] |  |  |  |
  Day 7: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
  Day 7 | 6 [4 to 6] |  |  |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 6 | 23 | 0 | 0
  Day 9 |  |  | 6 [6 to 8] | 4 [1 to 6] |  |
  Day 11: number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 11
  Day 11 |  | 6 [4 to 6] |  |  |  | 6 [4 to 12]
  Day 15: number analyzed (Participants) | 0 | 0 | 5 | 0 | 0 | 0
  Day 15 |  |  | 6 [4 to 8] |  |  |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 0
  Day 16 |  |  |  |  | 4 [2 to 8] |
  Day 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  Day 17 |  |  |  |  |  | 4 [2 to 6]
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0
  Day 22 |  |  |  |  | 4 [4 to 8] |
  Day 41: number analyzed (Participants) | 0 | 0 | 0 | 22 | 0 | 0
  Day 41 |  |  |  | 4 [4 to 8] |  |

22. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies to MEDI0382 (Cohorts 1, 2, 3, 4, 5, and 6)
Time Frame: Day 1 up to 7-14 days post-last dose of MEDI0382 for all cohorts (Approximately 60 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25 | 5 | 11 | 5 | 12
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Percent Change From Baseline in Insulin AUC0-4h After MMT to EOT (Cohorts 1, 2, 3, 4, 5, and 6)
Description: as for outcome 3
Time Frame: 0 minutes before; and 15, 30, 45, 60, 90, 120, 180, and 240 minutes post SMI on Baseline (Day -1) and EOT (Day 7 for Cohort 1; Day 11 for Cohort 2; Day 15 for Cohort 3; Day 41 for Cohort 4; Day 22 for Cohort 5; and Day 17 for Cohort 6)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25 | 5 | 11 | 5 | 12
Percent change | 10.83 (21.33) | -9.37 (29.17) | -3.67 (13.76) | 36.32 (35.21) | -20.43 (68.82) | -17.47 (38.84) | -8.63 (32.33) | -1.17 (44.20) | -17.70 (16.47) | 1.01 (31.00) | -8.18 (28.34) | -7.72 (37.03)

24. Secondary Outcome: Percent Change From Baseline in Proinsulin AUC0-4h After MMT to EOT (Cohorts 1, 2, 3, and 4)
Description: as for outcome 3
Time Frame: 0 minutes before; and 15, 30, 45, 60, 90, 120, 180, and 240 minutes post SMI on Baseline (Day -1) and EOT (Day 7 for Cohort 1; Day 11 for Cohort 2; Day 15 for Cohort 3; Day 41 for Cohort 4)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25
Percent change | -3.27 (38.92) | -52.10 (36.29) | -33.13 (40.07) | -36.77 (19.62) | 81.27 (77.21) | -54.13 (26.40) | -29.72 (31.13) | -47.93 (22.12)

25. Secondary Outcome: Percent Change From Baseline in C-peptide AUC0-4h After MMT to EOT (Cohorts 1, 2, 3, and 4)
Description: as for outcome 3
Time Frame: as for outcome 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25
Percent change | 10.17 (5.05) | -3.82 (21.29) | -1.43 (6.02) | 39.78 (32.88) | 79.37 (91.56) | -9.07 (27.27) | 8.08 (32.12) | 15.66 (42.35)

26. Secondary Outcome: Percent Change From Baseline in Incretin AUC0-4h After MMT to EOT (Cohorts 1, 2, 3, and 4)
Description: Mixes-meal test involved consumption of a standardized meal (nutritional supplement containing the components of fat, carbohydrate and protein, which make up a standard MMT) within 5 minutes, and timed serial blood samples were obtained for measurement of glucose and parameters related to glucose metabolism just before and 4 hrs after consumption of the standardized meal (with no additional food intake during this time). Incretins included glucagon-like peptide-1 (GLP-1; active and inactive both), glucagon, and gastric inhibitory peptide (GIP).
Time Frame: as for outcome 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3 | 7 | 26 | 25
Percent change
  GLP-1, Active: Change at EOT: number analyzed (Participants) | 2 | 6 | 3 | 6 | 3 | 5 | 24 | 19
  GLP-1, Active: Change at EOT | 8.30 (13.15) | -33.67 (16.84) | -10.40 (10.47) | -50.45 (12.30) | -2.87 (20.32) | -40.36 (26.90) | 1.63 (26.43) | -49.73 (22.88)
  GLP-1, Inactive: Change at EOT: number analyzed (Participants) | 1 | 1 | 1 | 3 | 2 | 3 | 14 | 8
  GLP-1, Inactive: Change at EOT | -20.30 (NA) — Standard deviation (SD) data not applicable as only one participant was evaluable for the specified parameter. | 0.70 (NA) — SD data not applicable as only one participant was evaluable for the specified parameter. | -22.90 (NA) — SD data not applicable as only one participant was evaluable for the specified parameter. | -10.93 (22.36) | 1.75 (29.20) | -8.07 (11.30) | 3.99 (29.59) | -28.85 (16.73)
  Glucagon: Change at EOT: number analyzed (Participants) | 2 | 4 | 3 | 5 | 3 | 2 | 18 | 12
  Glucagon: Change at EOT | -13.85 (18.60) | -20.25 (25.45) | -17.53 (19.46) | -38.12 (16.33) | -18.73 (21.59) | -3.05 (36.56) | -1.76 (21.47) | -30.17 (25.56)
  GIP: Change at EOT: number analyzed (Participants) | 2 | 2 | 2 | 5 | 2 | 5 | 17 | 12
  GIP: Change at EOT | 18.00 (2.83) | -46.50 (14.85) | 4.10 (24.61) | -27.08 (25.03) | -6.30 (7.35) | -21.34 (39.48) | -6.60 (19.43) | -37.38 (23.14)

ADVERSE EVENTS:
Time Frame: From Day 1 to follow-up period (28 days after the last study dose for each cohort [approximately 60 days])
Groups:
- Cohort 3: MEDI0382 200 mcg: Participants received MEDI0382 100 mcg SC once daily for at least 4 days (Day 1 to Day 4); thereafter, an up titrated dose of MEDI0382 150 mcg SC once daily for 4 days (Day 5 to Day 8); followed by second up titrated dose of MEDI0382 200 mcg SC once daily for 7 days (Day 9 to Day 15). )
Arm/Group | Cohort 1: Placebo | Cohort 1: MEDI0382 100 mcg | Cohort 2: Placebo | Cohort 2: MEDI0382 150 mcg | Cohort 3: Placebo | Cohort 3: MEDI0382 200 mcg | Cohort 4: Placebo | Cohort 4: MEDI0382 200 mcg | Cohort 5: Placebo | Cohort 5: MEDI0382 300 mcg | Cohort 6: Placebo | Cohort 6: MEDI0382 300 mcg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/6 | 0/3 | 0/7 | 0/26 | 0/25 | 0/5 | 0/11 | 0/5 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/6 | 0/3 | 1/7 | 1/26 | 0/25 | 0/5 | 0/11 | 0/5 | 0/12
Other Adverse Events (participants affected / at risk) | 2/3 | 6/6 | 3/3 | 5/6 | 3/3 | 7/7 | 23/26 | 22/25 | 4/5 | 10/11 | 2/5 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (N=3) | Cohort 1: MEDI0382 100 mcg (N=6) | Cohort 2: Placebo (N=3) | Cohort 2: MEDI0382 150 mcg (N=6) | Cohort 3: Placebo (N=3) | Cohort 3: MEDI0382 200 mcg (N=7) | Cohort 4: Placebo (N=26) | Cohort 4: MEDI0382 200 mcg (N=25) | Cohort 5: Placebo (N=5) | Cohort 5: MEDI0382 300 mcg (N=11) | Cohort 6: Placebo (N=5) | Cohort 6: MEDI0382 300 mcg (N=12)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (N=3) | Cohort 1: MEDI0382 100 mcg (N=6) | Cohort 2: Placebo (N=3) | Cohort 2: MEDI0382 150 mcg (N=6) | Cohort 3: Placebo (N=3) | Cohort 3: MEDI0382 200 mcg (N=7) | Cohort 4: Placebo (N=26) | Cohort 4: MEDI0382 200 mcg (N=25) | Cohort 5: Placebo (N=5) | Cohort 5: MEDI0382 300 mcg (N=11) | Cohort 6: Placebo (N=5) | Cohort 6: MEDI0382 300 mcg (N=12)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (7) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (9) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (5) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (8) | 1 (2) | 3 (4) | 4 (6) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 7 (7) | 0 (0) | 4 (7) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 3 (4) | 5 (7) | 13 (39) | 1 (2) | 3 (6) | 0 (0) | 5 (7)
Pancreatolithiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (8) | 0 (0) | 8 (40) | 0 (0) | 3 (9) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site erosion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site erythema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Medical device site injury (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic oedema (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram st segment depression (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 6 (6) | 0 (0) | 5 (5) | 1 (1) | 4 (4) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 4 (6) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (6) | 4 (6) | 2 (6) | 9 (10) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal mucosal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT02548585/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT02548585/SAP_001.pdf